CLINICAL TRIAL: NCT04802629
Title: Influence of Fetal Haemoglobin on Cerebral and Peripheral Oxygenation in Term and Preterm Neonates During the First Two Weeks After Birth Measured by Near Infrared Spectroscopy- a Prospective Observational Pilot Study
Brief Title: Fetal Haemoglobin and Cerebral and Peripheral Oxygenation.
Acronym: HbFIN
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: HbF Version 1.3
Record Dates: First submitted 2021-03-15; First posted 2021-03-17 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Preterm Birth; Oxygen Toxicity; Fetal Hemoglobin
Keywords: Fetal hemoglobin; preterm neonate; term neonate; near-infrared spectroscopy; cerebral oxygenation; peripheral oxygenation; fractional tissue oxygen extraction
MeSH Terms: conditions — Premature Birth; beta-Thalassemia | interventions — Spectroscopy, Near-Infrared

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Weeks
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Term neonates: ≥ 37+0 weeks of gestation
  Interventions: Device: Near-infrared spectroscopy
- Preterm neonates: ≤ 36+6 weeks of gestation
  Interventions: Device: Near-infrared spectroscopy

INTERVENTIONS:
Device: Near-infrared spectroscopy — For NIRS measurements the t-NIRS 1 and NIRO 200 NX (Hamamatsu, Japan) will be used. A cerebral sensor will be placed and fixed with a CPAP (Continuous Positive Airway Pressure) cap on the left forehead and a peripheral sensor on the right forearm. Duration of measurement will be two hours.

SUMMARY:
The aim of this study is to investigate the relationship between cerebral and peripheral oxygenation and oxygen extraction, as measured by NIRS (near-infrared spectroscopy ), and the FHbF (fraction of fetal hemoglobin) and absolute HbF (fetal hemoglobin) concentration in postnatal conditions in term and preterm neonates.

DETAILED DESCRIPTION:
During gestation the main fetal oxygen carrier is fetal hemoglobin (HbF). HbF exhibits a significantly higher affinity for oxygen when compared to adult hemoglobin (HbA), which makes it more suitable for oxygen extraction at the lower partial oxygen pressures in utero. Although the regulation of HbF expression is determined developmentally, recent studies report a respectable variation in the fraction of HbF in neonates.

Such data suggest that the differences in HbF expression could affect end-tissue oxygenation in neonates.

The methodology for measuring oxygen saturation and extraction in cerebral and peripheral tissues of neonates using the near-infrared spectroscopy (NIRS) has been well practiced in our study group. However, the method has not yet been used to investigate whether the fraction of fetal hemoglobin (FHbF) plays a significant role in cerebral and peripheral oxygenation in neonates.

The aim of this study is to investigate the relationship between cerebral and peripheral oxygenation and oxygen extraction, as measured by NIRS, and the FHbF and absolute HbF concentration in postnatal conditions in term and preterm neonates.

ELIGIBILITY:
Inclusion Criteria:

* Term and preterm neonates admitted to the neonatal intensive care unit (NICU)
* Decision to conduct full life support
* Written informed consent

Exclusion Criteria:

* No decision to conduct full life support
* No written informed consent
* Congenital malformations
* Family history of haemoglobinopathies (e.g. sickle cell anaemia, thalassaemia)

Ages: 2 Days to 3 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Preterm neonates (≤ 36+6 weeks of gestation) and term neonates (≥ 37+0 weeks of gestation) admitted to the NICU.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-06-08 (Actual); Primary Completion 2024-03-22 (Actual); Study Completion 2024-03-22 (Actual)

PRIMARY OUTCOMES:
FHbF (%) | First two weeks after birth
  Fraction of fetal hemoglobin in percentage
HbF (g/dL) | First two weeks after birth
  Fetal hemoglobin concentration in g/dL
Change of cTOI | at specific time points (2nd-3rd 6th-8th, 12th-14th day after birth)
  cerebral tissue oxygenation index (cTOI)
Change of pTOI | at specific time points (2nd-3rd 6th-8th, 12th-14th day after birth)
  peripheral tissue oxygenation index (pTOI)
Change of cFTOE | at specific time points (2nd-3rd 6th-8th, 12th-14th day after birth)
  cerebral fractional tissue oxygen extraction (cFTOE)
Change of pFTOE | at specific time points (2nd-3rd 6th-8th, 12th-14th day after birth)
  peripheral fractional tissue oxygen extraction (pFTOE)

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Pichler, Prof, Principal Investigator — Medical University of Graz
Locations (1):
- Department of Pediatrics, Division of Neonatology, Medical University of Graz, Graz, Styria, Austria

IPD SHARING:
Plan to Share IPD: Undecided